CLINICAL TRIAL: NCT02580032
Title: Validation of Two Measures for Growth Hormone Deficiency in Children, the Treatment Related Impact Measure of Childhood Growth Hormone Deficiency (TRIM-CGHD) and the Treatment Burden Measure of Childhood Growth Hormone Deficiency (TB-CGHD)
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8640-4231; U1111-1168-7911 (Other: WHO)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Growth Disorder; Growth Hormone Deficiency in Children
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Child Treatment Naïve group (Group A): Pre-pubertal boy or girl, ages of 9 to 13 years with a confirmed diagnosis of GHD prior to enrolment as determined by one GH stimulation test, defined as a peak GH level of equal or below 7.0 ng/ml.
  Interventions: Other: No treatment given
- Child Maintenance group (Group B): Pre-pubertal boy or girl, ages of 9 to 13 years with a confirmed diagnosis of GHD prior to enrolment as determined by one GH stimulation test, defined as a peak GH level of equal or below 10.0 ng/ml who have been taking prescription treatment for GHD for 6 months or more.
  Interventions: Other: No treatment given
- Parent Treatment Naïve group (Group C): Parents/guardians, who live with a pre-pubertal boy or girl, age 4 to 9 years with a confirmed diagnosis of GHD prior to enrolment as determined by one GH stimulation test, defined as a peak GH level of below or equal to 7.0 ng/ml.
  Interventions: Other: No treatment given
- Parent Maintenance group (Group D): Parents/guardians, who live with a pre-pubertal boy or girl, age 4 to 9 years with a confirmed diagnosis of GHD prior to enrolment as determined by one GH stimulation test, defined as a peak GH level of below or equal to 10.0 ng/ml who have been taking prescription treatment for GHD for 6 months or more.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given.

SUMMARY:
This study is conducted in Europe and the United States of America (USA). The aim of the study is to validate two measures for growth hormone deficiency in children, the Treatment Related Impact Measure of Childhood Growth Hormone Deficiency (TRIM-CGHD) and the Treatment Burden Measure of Childhood Growth Hormone Deficiency (TB-CGHD).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Child population - treatment näive:
* Confirmed diagnosis of Growth Hormone Deficiency (GHD) prior to enrolment as determined by a Growth Hormone (GH) stimulation test, defined as a peak GH level of 7.0 ng/ml or less. The GH stimulation test will be according to local clinical standards
* Pre pubertal children age 9 to less than 13 years at enrolment
* No prior exposure to GH therapy (GH-treatment naïve)
* Annualized height velocity (HV) below the 25th percentile for Chronological Age (CA) (HV less than -0.7 SD scores) and sex according to the standards of Prader et al (1989)
* Body Mass Index (BMI) percentile greater than 5th and below 95th percentile according to Centers for Disease Control and Prevention (CDC) BMI-for-age growth charts
* Child population - maintenance patients:
* Confirmed diagnosis of GHD prior to enrolment as determined by a GH stimulation test, defined as a peak GH level of 10.0 ng/ml or less. The GH stimulation test will be according to local clinical standards
* Pre pubertal children age 9 to less than 13 years at enrolment
* Body Mass Index (BMI) percentile greater than 5th and below 95th percentile according to Centers for Disease Control and Prevention (CDC) BMI-for-age growth charts
* Parent/Guardian population - treatment näive:
* Parent/Guardian of child with a confirmed diagnosis of GHD prior to enrolment as determined by a GH stimulation test, defined as a peak GH level of 7.0 ng/ml or less. The GH stimulation test will be according to local clinical standards
* Parent/Guardian of pre pubertal child age 4 to less than 9 years at enrolment
* Parent/Guardian of child with no prior exposure to GH therapy (GH-treatment naïve)
* Parent/Guardian of child with annualized height velocity (HV) below the 25th percentile for CA (HV less than -0.7 SD scores) and sex according to the standards of Prader et al (1989)
* Parent/Guardian of child with Body Mass Index (BMI) percentile greater than 5th and below 95th percentile according to Centers for Disease Control and Prevention (CDC) BMI-for-age growth charts
* Parent/Guardian living in the same residence as the child at least 50% of the time
* Parent/Guardian population - maintenance patients:
* Parent/Guardian of child with confirmed diagnosis of GHD prior to enrolment as determined by a GH stimulation test, defined as a peak GH level of 10.0 ng/ml or less. The GH stimulation test will be according to local clinical standards
* Parent/Guardian of pre pubertal child age 4 to less than 9 years at enrolment
* Parent/Guardian of child with Body Mass Index (BMI) percentile greater than 5th and below 95th percentile according to Centers for Disease Control and Prevention (CDC) BMI-for-age growth charts
* Parent/Guardian living in the same residence as the child at least 50% of the time Exclusion Criteria:
* Child population - treatment näive and maintenance patients:
* Any clinically significant abnormality likely to affect growth or the ability to evaluate growth:
* a) Chromosomal abnormalities and medical "syndromes", e.g. but not limited to Turner's syndrome, Laron syndrome, Noonan syndrome, or absence of GH receptors
* b) Congenital abnormalities (causing skeletal abnormalities), e.g. but not limited to Russell-Silver Syndrome, skeletal dysplasia's
* c) Significant spinal abnormalities including scoliosis, kyphosis and spina bifida variants - Children born small for gestational age (SGA - birth weight and/or birth length less than -2 SD for gestational age)
* Children diagnosed with diabetes mellitus or fasting blood glucose greater than or equal to 126 mg/dl (7.0 mmol/L), or HbA1c greater than or equal to 6.5% at enrolment
* Current inflammatory diseases (e.g. but not limited to arthritis, inflammatory bowel diseases) requiring systemic corticosteroid treatment or glucocorticoids treatment for longer than 2 weeks within the last 3 months prior to enrolment
* Children requiring glucocorticoid therapy (e.g. asthma) who are taking a dose of greater than 400 µg/day of inhaled budesonide or equivalents for longer than 1 month the year prior to enrolment
* Concomitant administration of other treatments that may have an effect on growth, e.g. but not limited to anabolic steroids and methylphenidate for attention deficit hyperactivity disorder (ADHD). Hormone replacement therapies (thyroxin, hydrocortisone, desmopressin) are allowed for inclusion
* Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* The subject and/or the parent/Legally Acceptable Representative (LAR) are likely to be non-compliant in respect to trial conduct, as judged by the investigator
* Parent/Guardian population - treatment näive and maintenance patients:
* Parent/Guardian of child with any clinically significant abnormality likely to affect growth or the ability to evaluate growth:
* a) Chromosomal abnormalities and medical "syndromes", e.g. but not limited to Turner's syndrome, Laron syndrome, Noonan syndrome, or absence of GH receptors
* b) Congenital abnormalities (causing skeletal abnormalities), e.g. but not limited to Russell-Silver Syndrome, skeletal dysplasia's
* c) Significant spinal abnormalities including scoliosis, kyphosis and spina bifida variants - Parent/Guardian of child born small for gestational age (SGA - birth weight and/or birth length less than -2 SD for gestational age)
* Parent/Guardian of child diagnosed with diabetes mellitus or fasting blood glucose greater than or equal to 126 mg/dl (7.0 mmol/L), or HbA1c greater than or equal to 6.5% at enrolment
* Parent/Guardian of child with current inflammatory diseases (e.g. but not limited to arthritis, inflammatory bowel diseases) requiring systemic corticosteroid treatment or glucocorticoids treatment for longer than 2 weeks within the last 3 months prior to enrolment
* Parent/Guardian of children requiring glucocorticoid therapy (e.g. asthma) who are taking a dose of greater than 400 µg/day of inhaled budesonide or equivalents for longer than 1 month the year prior to enrolment
* Parent/Guardian of child with concomitant administration of other treatments that may have an effect on growth, e.g. but not limited to anabolic steroids and methylphenidate for attention deficit hyperactivity disorder (ADHD). Hormone replacement therapies (thyroxin, hydrocortisone, desmopressin) are allowed for inclusion
* Parent/Guardian of child with any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* The subject and/or the parent/LAR are likely to be non-compliant in respect to trial conduct, as judged by the investigator

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The 2 populations (child and parent/guardian) will each be divided into a Treatment Naïve group and a Maintenance group.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Changes in CGI (Clinician Global Impression Scale) | After the physician scheduled MCID assessment visit (variable between week 3 and week 11) and week 12 follow-up visit after initiation of treatment

SECONDARY OUTCOMES:
Changes in PGI (Patient Global Impression Scale) | After the physician scheduled MCID assessment visit (variable between week 3 and week 11) and week 12 follow-up visit after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (27):
- United States (23):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Centennial, Colorado
  - Novo Nordisk Investigational Site, Wilmington, Delaware
  - Novo Nordisk Investigational Site, Margate, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Wheaton, Illinois
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Saint Paul, Minnesota
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Lebanon, New Hampshire
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Spring Valley, New York
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Dallas, Texas
- United Kingdom (4):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Derived] Brod M, Rasmussen MH, Alolga S, Beck JF, Bushnell DM, Lee KW, Maniatis A. Psychometric Validation of the Growth Hormone Deficiency-Child Treatment Burden Measure (GHD-CTB) and the Growth Hormone Deficiency-Parent Treatment Burden Measure (GHD-PTB). Pharmacoecon Open. 2023 Jan;7(1):121-138. doi: 10.1007/s41669-022-00373-z. Epub 2022 Oct 18. PMID 36255609
- [Derived] Brod M, Hojby Rasmussen M, Vad K, Alolga S, Bushnell DM, Bedoin J, Maniatis A. Psychometric Validation of the Growth Hormone Deficiency-Child Impact Measure (GHD-CIM). Pharmacoecon Open. 2021 Sep;5(3):505-518. doi: 10.1007/s41669-020-00252-5. Epub 2021 Jan 12. PMID 33433896
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com